CLINICAL TRIAL: NCT06437119
Title: A Randomized Double-blind Controlled Trial Study on the Antagonistic Effect of Composite Polyphenols on Health Damage Caused by Environmental Pollutants
Brief Title: The Antagonistic Effect of Composite Polyphenols on Health Damage Caused by Environmental Pollutants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Amway (China) Daily-Use Commodity Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Ruihua Dong, Associate Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB#2024-03-1102
Record Dates: First submitted 2024-05-21; First posted 2024-05-31 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Intestinal Functional Disorder; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Random numbers were generated using IBM SPSS Statistics 26.0, with the random seed set to the date of the day. Eligible participants were sorted based on the size of the generated random numbers, with the first 50% of the ranked list assigned to the placebo group and the last 50% assigned to the intervention group. Participants were allocated randomly in equal proportions, and the random list was validated by a statistician.
Who Masked: Participant, Investigator
Masking Description: The on-site implementation personnel and those responsible for coordinating the study only received the study number of the subjects, and were unaware of the intervention group allocation of the subjects. The subjects were also unaware of their intervention allocation. A copy of the sealed envelope of the non blinded study number for each subject is provided only to the study supervisor. Before the completion of data collection, the investigators and researchers kept the blind method for treatment allocation. All subjects were monitored in a double-blind way throughout the study period, and the subjects could not distinguish their own grouping by asking questions or from appearance and texture.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition supplement group (Experimental): The Composite polyphenols intervention agent includes extracts of licorice, sophora, wild cherry berry, dendrobium officinale, and pomegranate. They should be taken three times a day, one pack at a time, brewed and dissolved in warm water, and taken with meals or after meals.
  Interventions: Dietary Supplement: Compound plant nutrients
- placebo group (Placebo Comparator): A placebo with an indistinguishable appearance and color. 3 times a day, 1 pack at a time, dissolve in warm water and take with meals or after meals.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Compound plant nutrients — The compound plant nutrients include extracts of licorice, sophora, wild cherry berry, dendrobium officinale, and pomegranate.
  Arms: Nutrition supplement group
Dietary Supplement: placebo — A placebo with an indistinguishable appearance and color.
  Arms: placebo group

SUMMARY:
The study attempts to conduct randomized controlled trials to understand whether daily exposure to environmental pollutants can cause harm to human health, explore whether the intake of composite polyphenols can alleviate potential health hazards caused by environmental pollutants, and provide scientific basis for the prevention and treatment of health hazards caused by environmental pollutant exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18-65 years; 2. Body mass index (BMI) < 35 kg/m²; 3. On-campus residence for one year and no need to leave the province during the trial period; 4. Agreeing to and signing the informed consent form.

Exclusion Criteria:

1.Documented diagnosis of congenital or acquired immunodeficiency disorders, allergic diseases, gastrointestinal pathologies, or other acute/chronic conditions requiring therapeutic intervention; 2.Administration of immunosuppressive agents, antibiotics, probiotics, prebiotics, synbiotics, or gastrointestinal motility-active medications within three months prior to the trial; 3.Consumption of nutritional supplements within three months preceding the study; 4.Underlying disease, including hypertension or diabetes mellitus; 5.Habitual substance use (tobacco smoking or alcohol consumption); 6.Influenza vaccination within 12 months prior to the trial; 7.pregnancy or lactation status; 8.Body weight fluctuation exceeding 5% within three months before the study; 9.Concurrent or planned enrollment in alternative clinical investigations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Fecal microplastics (MPs) levels as assessed by Py-GC/MS | up to 2 months
  Py-GC/MS method for detecting microplastic (MPs) levels in feces of research subjects. The concentration of fecal microplastics will be reported in units of μ g/g dry weight (μ g/g dw)
Fecal metagenomic sequencing as sequenced using the Illumina NovaSeq/HiSeq Xten platform | up to 2 months
  DNA was extracted from fecal samples using the FastPure Stool DNA Isolation Kit (Magnetic bead) (MJYH, Shanghai, China). The DNA fragments were amplified via bridge PCR and sequenced using the Illumina NovaSeq/HiSeq Xten platform (Illumina, USA). Raw data were processed using Fastp and BWA software for quality control and removal of host DNA sequences. The abundance of genes in each sample was described using RPKM.
Blood Metabolomics as assessed by UPLC-TripleTOF | About 2 months
  The pretreated samples were analyzed using an Ultra-high Performance Liquid Chromatography with quadrupole time-of-flight mass spectrometry (UPLC-TripleTOF) system (AB SCIEX). The samples were separated using a BEH C18 chromatography column (100 mm*2.1 mm i.d., 1.8 µm) and detected via mass spectrometry. The mass spectrometry signal was acquired in positive and negative ion scanning modes, with a mass-to-charge ratio (m/z) range of 50-1000. Raw data were imported into the Progenesis QI software (Waters Corporation, Milford, USA) for processing, generating a data matrix containing retention time, m/z, and peak intensity. The MS and MS/MS spectra were matched with the HMDB (http://www.hmdb.ca/) and Metlin (https://metlin.scripps.edu/) databases to identify metabolites.
Inflammatory cytokines as assesed by Luminex technology | About 2 months
  The levels of 10 inflammatory cytokines in blood plasma samples were detected using Luminex technology, including IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, TNF-α, and IFN-γ. Inflammatory cytokine indicators are described in pg/ml units.
Blood glucose indicators as assessed by the Hitachi 7180 fully automatic biochemical analyzer | About 2 months
  Using the Hitachi 7180 fully automatic biochemical analyzer to measure glucose (glycated serum protein, GSP; glucose, GLU) indicators. Blood glucose indicators are described in mmol/l units.
Blood lipid indicators as assessed by the Hitachi 7180 fully automatic biochemical analyzer | about 2 months
  Using the Hitachi 7180 fully automatic biochemical analyzer to measure lipid (total cholesterol, CHO; triglycerides, TG; high-density lipoprotein cholesterol, HDL; low-density lipoprotein cholesterol, LDL) indicators. Blood lipid indicators are described in mmol/l units.
Routine blood examination as assessed by the Dima DH36X fully automatic blood cell analyzer | About 1 months
  Using the Dima DH36X fully automatic blood cell analyzer for routine blood examination (three-part differential). We measured the white blood cell count (WBC), lymphocyte count (LYM), monocyte count (MXD), and neutrophil count (NEU) in the blood routine and reported them in units of 10 * 9 cells/L

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Dong, Principal Investigator — School of Public Health，Fudan University
Locations (1):
- School of Public Health, Fudan University, Shanghai, Xuhui, China

IPD SHARING:
Plan to Share IPD: No